CLINICAL TRIAL: NCT04091152
Title: Usability Assessment of a Tablet PC Designed for Old Patients: the "Ardoiz" Tikeasy Tablet.
Brief Title: TIKeasy TAblet satisfaCtion (TikTac)
Acronym: TikTac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019/41
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Old Age; Debility; Satisfaction
Keywords: old poeple; elderly; usability; ergonomy; tablet PC
MeSH Terms: conditions — Frailty; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- old patients: Patient will freely use "Ardoiz" during their hospitalisation for a maximum of 9 days.
  After this use, a survey concerning the usability of "Ardoiz" will be administered to the patient, before their discharge from hospital.
  Interventions: Other: usability assessment
- relatives / unformal caregivers: Unformal caregivers will freely use "Ardoiz" during the hospitalization of their relatives and a maximum of 9 days.
  After this use, a survey concerning the usability of "Ardoiz" will be administered to the unformal caregivers, before the discharge of their hospitalized relatives from hospital.
  Interventions: Other: usability assessment
- profesionnal caregivers: After the inclusion of all expected patients and relatives, a survey concerning the usability of "Ardoiz" will be administered to professional caregivers.
  Interventions: Other: usability assessment

INTERVENTIONS:
Other: usability assessment — Usability of "ardoiz" will be assesse using a validated usability questionnary

SUMMARY:
In the last ten years, gerontechnology is becoming an increasing topic in geriatric medicine. Nevertheless, there are still few studies assessing the usability of technologies in old patients, especially when they are hospitalized. Moreover, it has been shown that new technologies could be a source of ageism, thence the importance of involving the old people in the development of these technologies.

Tik easy is a subsidiary of La Poste Company. Tik easy as designed a new tablet PC for old people. Research tends to show that the use of tablet PC can promote health and well-aging, and delay cognitive decline. In this study, we want to give a free access to "Ardoiz", the tablet PC designed by Tik easy, for old patients hospitalized in a geriatric acute care unit. The "Ardoiz" tablet PC allows to:

* Maintain the family and social bond (send and receive messages, share photos and videos, call remotely between the patient and his family)
* Discovering the Internet at his own pace (browse the Internet with daily updated contents such as news, content on cooking, music, etc.).
* Prevent cognitive aging (stimulate cognitive abilities with the DYNSEO games).
* Facilitate online administrative procedures.

DETAILED DESCRIPTION:
The "Ardoiz" tablet PC will be given to old patients hospitalized in the acute care geriatric unit of the university hospital of Angers. Patients and their relatives will have a free access to "Ardoiz" during their hospitalisation. The maximum duration of use will be 9 days. After the using period, a survey will be proposed to the patients and their relatives. This survey include questions concerning usability (using the validated SUS questionnaire), ergonomics (using non validated specific questionnaire with closed questions oriented on "Ardoiz" device), satisfaction (general and specific questions using non validated questionnaire with forced choice Likert scale in 4 points and closed questions). After recruiting all expected patients and relatives; the survey will also be submitted to the professional caregivers of the unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients :

  * Aged 65 years old and over
  * To be hospitalised in geriatric medicine department of Angers University Hospital
* Caregivers:

  * Family members or relatives
  * Aged 18 years old and over
* Healthcare team :

  * geriatric medicine department's staff of Angers University Hospital
  * Aged 18 years old and over

Exclusion Criteria:

* Patients :

  * Existence of a delirium revealed by the Confusion Assessment Method
  * To be under legal protection
* Refusal of participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited during their hospitalisation in geriatric medicine. Relatives / unformal caregivers are recruited during the hospitalisation of patients in geriatric medicine.
  Professionnal caregivers are recruited in the acute care geriatric unit.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-09-16 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
Usability of the Ardoiz® tablet PC | During the 48 hours before the discharge of the hospital
  The usability will be assessed using the validated System Usability Scale (SUS). The mean score obtained by users will be calculated. "Ardoiz" will be considered as usable if the mean score on the SUS is equal or over 70 on 100.

SECONDARY OUTCOMES:
Satisfaction of the users following the use of the Ardoiz® tablet PC. | During the 48 hours before the discharge of the hospital
  The satisfaction will be assessed using a non-validated satisfaction questionnaire based on a forced choice Likert scale in 4 points from 1 to 4. The mean score obtained by users will be used. Users will be considered as satisfied if the mean score is over 2 on 4.
Frequency of use of the Ardoiz® tablet PC by elderly hospitalized patients. | During the 48 hours before the discharge of the hospital
  The frequency of use will be described using a non-validated questionnary based on 4 closed questions.
Most appreciated ergonomic elements for the users | During the 48 hours before the discharge of the hospital
  The ergonomic elements will be assessed using a single choice closed liste of ergonomic elements. The most ergonomic elements will be ranked in descending order of citation by users.
Improvement areas regarding the ergonomics of the Ardoiz® tablet PC. | During the 48 hours before the discharge of the hospital
  The ergonomic elements will be assessed using a single choice closed liste of ergonomic elements. The less ergonomic elements will be ranked in descending order of citation by users.
Improvement areas regarding the functions of the Ardoiz® tablet PC. | During the 48 hours before the discharge of the hospital
  The satisfaction concerning functions of "Ardoiz" will be assessed using a single choice closed liste of functions. The less appreciated functions will be ranked in descending order of citation by users.

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Annweiler, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France